CLINICAL TRIAL: NCT02986542
Title: Comparison of Success Rates of Femoral Artery Catheterization for Newborns With In-plane and Out-of-plane Ultrasonography Techniques
Brief Title: Comparison of Success Rates of Femoral Artery Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ömer Faruk Boran, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 255
Record Dates: First submitted 2016-11-18; First posted 2016-12-08 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Disease; Electrolyte Disorder; Metabolic Disease; Sepsis
Keywords: newborns,femoral artery, catheterization
MeSH Terms: conditions — Lung Diseases; Metabolic Diseases; Sepsis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- USG with the in-plane technique (Active Comparator): Intervention: Femoral artery catheterization under USG guidance with the in-plane technique.Patients will have their femoral arterial lines inserted under the guidance of USG. The ultrasound equipment used is LOGIQ e GE medical system(China) CO.LTD
  Interventions: Procedure: Femoral artery catheterization
- USG with the out-of-plane technique (Active Comparator): Intervention: Under USG guidance femoral artery catheterization will be done with the probe placed for the out-of-plane technique. The ultrasound equipment used is LOGIQ e GE medical system(China) CO.LTD
  Interventions: Procedure: Femoral artery catheterization

INTERVENTIONS:
Procedure: Femoral artery catheterization — The intervention will be performed by a single experienced individual.

SUMMARY:
The use of USI has eased practical application of interventional procedures, and reduced complications and procedure durations. For vascular interventions with ultrasound imaging, short- or long-section imaging of vascular structures is performed. Both techniques have their own advantages and disadvantages.

This study aims to compare the success rates of femoral artery catheterization using both imaging techniques.

DETAILED DESCRIPTION:
The research will include newborns undergoing open heart surgery and patients requiring arterial monitoring in the neonatal intensive care unit. Eighty patients requiring femoral artery cannulation will be randomized with the closed envelope method and separated into two groups as USI with the in-plane technique (Group A) and USI with the out-of-plane technique (Group B). The intervention will be performed by a single experienced individual. The preparation duration, puncture duration, number of punctures, number of unsuccessful arterial punctures, development of hematoma and other complications will be recorded and the groups will be compared. If there are 3 unsuccessful attempts the procedure will be ended.1. Patients undergoing KVC surgery and patients requiring arterial catheterization in the neonatal intensive care unit (cases with pulmonary disease, electrolyte disorders, metabolic disease, or sepsis requiring frequent blood sampling) EXCLUSION CRITERIA FOR STUDY VOLUNTEERS

1. Local infection
2. Coagulopathy CLINICAL END-POINTS (MEASURED VARIABLES)

1. Distance of femoral artery to skin, distance of femoral artery to inguinal ligament, femoral artery diameter, femoral artery and vein location properties 2. Preparation duration, number of punctures, complications developing during the procedure

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing KVC surgery and patients requiring arterial catheterization in the neonatal intensive care unit (cases with pulmonary disease, electrolyte disorders, metabolic disease, or sepsis requiring frequent blood sampling

Exclusion Criteria:

1. Local infection
2. Coagulopathy

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03-25 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Femoral artery catheterization puncture duration | 1 - 5 minutes

SECONDARY OUTCOMES:
Number of Attempts | 5 minutes
Rate of Success of First Attempt | 1 - 5 minutes
Distance of femoral artery to skin | 1 - 5 minutes
  Distance of femoral artery to skin
Distance of femoral artery to inguinal ligament | 1 - 5 minutes
Femoral artery diameter | 1 - 5 minutes
Complications developing during the procedure | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Faruk Boran, Study Chair — Kahramanmaraş Üniversitesi
Locations (1):
- Kahramanmaraş Sütçü Imam Üniversity, Kahramanmaraş, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No